CLINICAL TRIAL: NCT05034757
Title: The Development of a Guidance of Combined Hyaluronate and Extracorporeal Shockwave Therapy (ESWT) for Non-calcific Rotator Cuff Lesions Without Complete Tear
Brief Title: The Development of a Guidance of Combined HA and ESWT for Non-calcific Rotator Cuff Lesions Without Complete Tear
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Jih-Yang Ko, Professor, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201900290B0A3
Record Dates: First submitted 2021-08-03; First posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Rotator Cuff Lesions
Keywords: HA; ESWT; non-calcific rotator cuff lesions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyaluronate (Experimental): HA injection
  Interventions: Other: HA only
- HA + ESWT (Experimental): HA + ESWT
  Interventions: Other: ESWT once; Other: ESWT twice

INTERVENTIONS:
Other: HA only — HA injection only
  Arms: Hyaluronate
Other: ESWT once — ESWT of the shoulder the patient will receives STORZ Extracorporeal Shock Wave Therapy 3000 impulses (each point) of shockwaves at 24kV (energy flux density, 0.32mJ/mm2) to the affected shoulder
  Arms: HA + ESWT
Other: ESWT twice — ESWT of the shoulder the patient will receives STORZ Extracorporeal Shock Wave Therapy 3000 impulses (each point) of shockwaves at 24kV (energy flux density, 0.32mJ/mm2) to the affected shoulder
  Arms: HA + ESWT

SUMMARY:
The rotator cuff lesions are common disorders of the shoulder joint and mainly caused by intrinsic degeneration and outlet impingement. The symptoms include pain, discomfort, weakness, range of motion limitation, and impingement. The initial treatment of rotator cuff lesions are non-surgical especially for non-full thickness tearing and include rehabilitation and medications given orally, topically, or parenterally. Although many patients with rotator cuff lesions or subacromial pain are treated with, and will respond to non- surgical treatment alone, surgical intervention with subacromial decompression and rotator cuff repair is often used as an early treatment choice or in recalcitrant cases. The indications for surgery are persistent and severe shoulder pain combined with functional restrictions that are resistant to conservative measures. However, the effectiveness of this procedure is still elusive. Some studies have compared decompression plus subacromial bursectomy with bursectomy alone and reported no significant difference in clinical outcome between groups.

In addition, arthroscopic subacromial decompression for shouled impingement was currently challenged because some high-quality prospective studies including that from Oxford university showed similar outcomes between surgical and non-surgical treatment. Therefore more efficient non-surgical treatments were needed for the rotator cuff lesions without complete tear.

The investigators have successfully treated non- calcific rotator cuff lesions without complete tearing with hyaluronate and published our data in J Shoulder Elbow surgery. Jun 19:557-63, 2010.

In the Phase III study, the investigators will perform three subacromial hyaluronate injections and zero to two sessions of extracorporeal shock wave therapy (ESWT) for these patients. The investigators hypothesize that through the actions of anti-inflammation, neovascularization and temporary cell permeability increment, a combined therapy of HA and ESWT may offer better therapeutic effects on the non-calcific rotator cuff lesion without complete tearing. The investigators will evaluate the treatment effects with Constant score and VAS scale and also check the changes or expressions of cytokines, growth factors, functional proteins, from the peripheral blood.

DETAILED DESCRIPTION:
The rotator cuff lesions are common disorders of the shoulder joint and mainly caused by intrinsic degeneration and outlet impingement. The symptoms include pain, discomfort, weakness, range of motion limitation, and impingement. The initial treatment of rotator cuff lesions are non-surgical especially for non-full thickness tearing and include rehabilitation and medications given orally, topically, or parenterally.

Although many patients with rotator cuff lesions or subacromial pain are treated with, and will respond to non- surgical treatment alone, surgical intervention with subacromial decompression and rotator cuff repair is often used as an early treatment choice or in recalcitrant cases. The indications for surgery are persistent and severe subacromial shoulder pain combined with functional restrictions that are resistant to conservative measures. However, the effectiveness and necessity of this procedure is still elusive. Some studies have compare decompression plus subacromial bursectomy with bursectomy alone and reported no significant difference in clinical outcome between groups.

In addition, arthroscopic subacromial decompression for shouled impingement was currently challenged because some high-quality prospective studies including that from Oxford university showed similar outcomes between surgical and non-surgical treatment. Therefore more efficient non-surgical treatments were needed for the rotator cuff lesions without complete tear.

The investigators have successfully treated non-calcific rotator cuff lesions without complete with hyaluronate and published our data in J Shoulder Elbow Surg. Jun 19:557-63,2010.

In the phase III study, the investigators will perform three subacromial hyaluronate injections and zero to two sessions of extracorporeal therapy (ESWT). The investigators hypothesize that through the actions of anti-inflammation, neovascularization and temporary cell permeability increment of ESWT, a combined therapy of HA and ESWT may offer better therapeutic effects on the non-calcific rotator cuff lesion without complete tearing. The investigators will evaluate the treatment effects with constant score and VAS, and also check the changesor expressions of cytokines, growth factors, functional protein, from the peripheral blood.

1. Acceptance criteria:

   The randomized, double-blind, placebo-controlled clinical study will involve 69 or more patients who have non-calcific rotator cuff lesions without complete tear. The inclusion criteria are (1) patients who have pain around the shoulder, a positive impingement sign, and a positive imaging diagnosis of rotator non-calcific cuff pathology without complete tear; (2) patients who do not respond to conservative therapy or rehabilitation for at least 3 months; and (3) patients age between 35 and 80 years, who sign the informed consent form. The investigators will exclude patients who have rheumatic diseases, glenohumeral osteoarthritis, full-thickness cuff tears, fractures, infections, or tumors; those who have received a subacromial injection within 3 weeks; and those who are pregnant or want to become pregnant.

   The sample size is calculated under the expectation of an improvement in the Constant score of 10 points, with an SD of 12 points in each group, and a power value of 0.8. For this study design, the minimal number of patients required in each group is 23, by use of an independent-samples t test. The intent-to-treat population is a fully randomized group of patients who have a baseline value (Constant score and VAS before treatment). The imaging diagnosis of a rotator cuff lesion is made by a musculoskeletal radiologist who has considerable experience in interpreting both magnetic resonance imaging (MRI) and sonographic results for shoulders. On the sonogram, hypoechoic thickening of the rotator cuff indicates tendinosis. Focal thinning or focal hypoechoic areas of discontinuity in the rotator cuff are suggestive of partial-thickness tearing. In cases of the hypoechoic gap extending through the entire rotator cuff, tendon retraction, or the absence of a visible rotator cuff, a full thickness tear is assumed to be present. On MRI, rotator cuff tendinosis is characterized by increased intratendinous signal intensity on T2-weighted images without tendon disruption. Partial-thickness tearing is characterized by the presence of focal hyperintense fluid or a fluid-like signal intensity that extended into the tendon on the T2-weighted images. A full thickness tear is diagnosed by the extension of hyperintense fluid or fluid-like signal intensity through the entire thickness of the interrupted rotator cuff tendon on T2-weighted images.
2. Experiment design and method Patients are then randomly into three groups and every patient receives three injections of HA along with ESWT treatment based on statistical randomization. For ESWT of the shoulder the patient will receive Storz Extracorporeal Shock Wave Therapy 3000 impulses (each point) of shockwaves at 24kV (energy flux density, 0.32mJ/mm2) to the affected shoulder. Treatments are performed on an outpatient basis. The areas of treatment (2 points) near the supraspinatus insertion is focused with a control guide on the machine, and surgical lubricant is placed on the skin in contact with the shockwave tube. The sham treatment entails use of the same device in which the shockwave generator is disconnected. The patients' vital signs and local discomfort are monitored throughout the course of treatment. The treated area is inspected for local swelling, ecchymosis, or hematoma immediately after the treatment. Our primary endpoint is the Constant Score improvement by 10 points and the treatment success is followed up to 1 year. The Constant score pain score and the range of shoulder motion are measured. Another kind of pain and pain that requires surgery is classified as a failure case, which is the secondary endpoint.
3. Rehabilitation including gentle flexion, abduction, internal rotation and external rotation exercises, pendulum exercises, and resistant exercises will be instructed and continued during the study period.

Patients will have a pain medication-free interval 2 days prior to each evaluation. After treatment and during follow-up, patients will be restricted to the use of a 750mg of acetaminophen per day for pain, in order to fascilitate usage and comparison of the medications among the patients. Follow-up examinations with range of motion, VAS and Constant score are performed independently by one of the coauthors, who is blinded to patient treatment status during the treatment course and at 1week, 1month, 3months, 6 months, and 12 months after treatment. Peripheral blood (10cc) will be collected during the treatment course and 1 week, 1 month and 3 month after treatment and shoulder MRI will be checked 12 months after treatment. Patients who have persistent shoulder discomfort may be advised to undergo surgical intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Pain around the shoulder, a positive impingement sign
2. Diagnosis of non-calcific rotator cuff pathology without complete tear
3. Do not respond to conservative therapy or rehabilitation for at least 3 months

Exclusion Criteria:

1. Rheumatic diseases
2. Glenohumeral osteoarthritis
3. Full-thickness cuff tears
4. Fractures
5. Infections
6. Tumors
7. Received a subacromial injection within 3 weeks
8. Pregnant or want to become pregnant.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2019-10-31 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Constant Score | measure and record during the treatment course.
  The Constant Score contains pain (15 points), activities of daily living (20 points), mobility (40 points), and strength (25 points). Improve the Constant Score by 10 points for treatment success. For monitoring the participants' recovery progress, will measure and record during the treatment course.
Constant Score | measure and record at 1 month after treatment.
  The Constant Score contains pain (15 points), activities of daily living (20 points), mobility (40 points), and strength (25 points). Improve the Constant Score by 10 points for treatment success. For monitoring the participants' recovery progress, will measure and record at 1 month after treatment.
Constant Score | measure and record at 3 months after treatment.
  The Constant Score contains pain (15 points), activities of daily living (20 points), mobility (40 points), and strength (25 points). Improve the Constant Score by 10 points for treatment success. For monitoring the participants' recovery progress, will measure and record at 3 months after treatment.
Constant Score | measure and record at 6 months after treatment.
  The Constant Score contains pain (15 points), activities of daily living (20 points), mobility (40 points), and strength (25 points). Improve the Constant Score by 10 points for treatment success. For monitoring the participants' recovery progress, will measure and record at 6 months after treatment.
Constant Score | measure and record at 12 months after treatment.
  The Constant Score contains pain (15 points), activities of daily living (20 points), mobility (40 points), and strength (25 points). Improve the Constant Score by 10 points for treatment success. For monitoring the participants' recovery progress, will measure and record at 12 months after treatment.
visual analog scale (VAS) | measure and record during the treatment course.
  Assess whether the pain level is reduced. The VAS with two endpoints representing 0 ('no pain') and 10 ('extreme pain'). For monitoring the patients' recovery progress, will measure and record during the treatment course.
visual analog scale (VAS) | measure and record at 1 month after treatment.
  Assess whether the pain level is reduced. The VAS with two endpoints representing 0 ('no pain') and 10 ('extreme pain'). For monitoring the patients' recovery progress, will measure and record at 1 month after treatment.
visual analog scale (VAS) | measure and record at 3 months after treatment.
  Assess whether the pain level is reduced. The VAS with two endpoints representing 0 ('no pain') and 10 ('extreme pain'). For monitoring the patients' recovery progress, will measure and record at 3 months after treatment.
visual analog scale (VAS) | measure and record at 6 months after treatment.
  Assess whether the pain level is reduced. The VAS with two endpoints representing 0 ('no pain') and 10 ('extreme pain'). For monitoring the patients' recovery progress, will measure and record at 6 months after treatment.
visual analog scale (VAS) | measure and record at 12 months after treatment.
  Assess whether the pain level is reduced. The VAS with two endpoints representing 0 ('no pain') and 10 ('extreme pain'). For monitoring the patients' recovery progress, will measure and record at 12 months after treatment.
Range of Motion (ROM) | measure and record during the treatment course.
  Assess whether the range of motion is increased. Measure the motions: abduction, elevation through flexion, external rotation and internal rotation. For monitoring the patients' recovery progress, will measure and record during the treatment course.
Range of Motion (ROM) | measure and record at 1 month after treatment.
  Assess whether the range of motion is increased. Measure the motions: abduction, elevation through flexion, external rotation and internal rotation. For monitoring the patients' recovery progress, will measure and record at 1 month after treatment.
Range of Motion (ROM) | measure and record at 3 months after treatment.
  Assess whether the range of motion is increased. Measure the motions: abduction, elevation through flexion, external rotation and internal rotation. For monitoring the patients' recovery progress, will measure and record at 3 months after treatment.
Range of Motion (ROM) | measure and record at 6 months after treatment.
  Assess whether the range of motion is increased. Measure the motions: abduction, elevation through flexion, external rotation and internal rotation. For monitoring the patients' recovery progress, will measure and record at 6 months after treatment.
Range of Motion (ROM) | measure and record at 12 months after treatment.
  Assess whether the range of motion is increased. Measure the motions: abduction, elevation through flexion, external rotation and internal rotation. For monitoring the patients' recovery progress, will measure and record at 12 months after treatment.
MRI | shoulder MRI will be checked 12 months after treatment
  Take shoulder MRI to compare the difference before and after treatment. The degeneration of the supraspic is graded as: grade 1 ≤ 1/3; 1/3 < grade 2 < 2/3; grade 3 ≥ 2/3.

CONTACTS AND LOCATIONS:
Overall Officials: Jih-Yang Ko, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Derived] Ko JY, Huang CC, Huang PH, Chen JW, Liao CY, Kuo SJ. Effects of supplementing extracorporeal shockwave therapy to hyaluronic acid injection among patients with rotator cuff lesions without complete tear: a prospective double-blinded randomized study. Int J Surg. 2024 Dec 1;110(12):7421-7433. doi: 10.1097/JS9.0000000000002063. PMID 39172722